CLINICAL TRIAL: NCT04094662
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled 14-week Study of DS-5565 in Chinese Patients With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DS5565-A-A315
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — mirogabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirogabalin (Experimental): Mirogabalin 15 mg, oral administration, Treatment period; 2-weeks titration and 12-weeks maintenance dose.
  Interventions: Drug: Mirogabalin
- Placebo (Placebo Comparator): Placebo (14-weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirogabalin — Mirogabalin tablets for oral administration
  Other Names: DS-5565
  Arms: Mirogabalin
Drug: Placebo — Matching placebo tablets for oral administration
  Arms: Placebo

SUMMARY:
Investigate the efficacy and safety of mirogabalin in Chinese participants with diabetic peripheral neuropathic pain in comparison to placebo.

DETAILED DESCRIPTION:
The primary objective is to compare change from baseline in weekly Average Daily Pain Score (ADPS) at Week 14 in Chinese patients with Diabetic Peripheral Neuropathic Pain (DPNP) receiving mirogabalin versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus at screening
* Painful distal symmetric polyneuropathy, diagnosed at least 6 months prior to screening (see Procedures manual for the Diagnosis of Diabetic Peripheral Neuropathy and Neurological Examination for details)

Exclusion Criteria:

* HbA1c (National Glycohemoglobin Standardization Program) > 10.0% at screening
* Uncontrolled blood glucose within 1 month prior to screening, at screening or randomization
* Other severe pain at screening or randomization, unrelated to DPN, that may confound the assessment of DPNP
* Neurologic disorders at screening or randomization, unrelated to DPN, that may confound the assessment of DPNP
* Major psychiatric disorders at screening or randomization
* Creatinine clearance (using the Cockcroft-Gault equation) < 60 mL/min at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Average Daily Pain Score (ADPS) | Baseline to Week 14
  The pain scores on a scale of 0-10, where 0 = no pain and 10 = the worst possible pain. The weekly ADPS is based on participants daily pain scores.

SECONDARY OUTCOMES:
ADPS responder rate | at Week 14
  Ratio of Participants Responding to Treatment, as Measured by Average Daily Pain Score (ADPS) Reduction from Baseline. The ADPS is used to determine categorical response rates.
Pain Intensity Score Using the Short-Form McGill Pain Questionnaire (SF-MPQ): Visual Analog Scale (VAS) | at Week 14
  The VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.
Patient Global Impression of Change | at Week 14
  Participants rate their overall impression of how the present pain compares to baseline using a 7-point scale, where 1 = very much improved and 7 = very much worse. Patient Global Impression of Change scores are used to determine categorical responder rates.
Average Daily Sleep Interference score (ADSIS) | at Week 14
  The sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. The weekly ADSIS is based on participants daily sleep interference scores.
Medical Outcome Study (MOS) sleep scale | at Week 14
  Participants rate their sleep quality during the past 4 weeks in three parts of the questionnaire:
  Part 1 - The participants rate the average time required to fall asleep, 0-15 minutes = 1, 16-30 minutes = 2, 31-45 minutes = 3, 46-60 minutes = 4, More than 60 minutes = 5.
  Part 2 - The participants give the number of hours per night for the average hours of sleep per night.
  Part 3 - The participants using a score of 1 (all of the time) to 5 (none of the time) to rate their sleep disturbance in the following areas: difficulty in falling asleep or remaining asleep, difficulty in staying awake during the day, difficulty in breathing, and snoring during sleep.
Five Level EuroQol-5D (EQ-5D) version | at Week 14
  Participants rate their Quality of Life in the following dimensions: mobility (5-point scale), self-care (5-point scale), usual activities (5-point scale), pain/discomfort (5-point scale), and anxiety/depression(5-point scale) that are combined into an overall health utilities index. Participants also rate their perception of overall health using VAS, with zero indicating worst health and 100 representing best imaginable health.

OTHER OUTCOMES:
Actigraphy signal collected from a wrist-worn medical-grade sensor | at Week 14
  Result of physical activity during waking hours and participants' sleep will be evaluated to explore a relationship between participants reported outcomes and actigraphy signal collected from a wrist-worn medical-grade sensor (ActiGraph GT9X Link). Only participants who signed a separate informed consent form for wearing medical-grade sensor will be included in this evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (40):
- China (40):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Special Medical Center of Chinese PLA Rocket Force, Beijing
  - Beijing PingGu Hospital, Beijing
  - Cangzhou Central Hospital, Cangzhou
  - Jilin Province People's Hospital, Changchun
  - The First Hospital of Changsha, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Peace Hospital Affiliated to Changzhi Medical College, Changzhi
  - West China Hospital, Sichuan University, Chengdu
  - The Fourth People's Hospital of Chongqing, Chongqing
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - Foshan First People's Hospital, Foshan
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - Guizhou Provincial People's Hospital, Guizhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jiaxing Second Hospital, Jiaxing
  - Jilin Central General Hospital, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jingzhou
  - Yunnan First People's Hospital, Kunming
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Luoyang Central Hospital Affiliated to Zhengzhou University, Luoyang
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai Huashan Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Yangpu Hospital,Tongji University, Shanghai
  - Shanghai Pudong Hospital, Shanghai
  - Central Hospital of Minhang District Shanghai, Shanghai
  - Siping Central Hospital, Siping
  - The First Hospital of Shanxi Medical University, Taiyuan
  - The Second Hospital of Tianjin Medical University, Tianjin
  - The 2nd Affiliated Hospital of The 2nd School of Medicine, Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University (Hubei General Hospital), Wuhan
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zigong Fourth People's Hospital, Zigong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Guo X, Yu Y, Zhang Y, Sun L, Li Y, Song B, Hang L, Baba M, Wasaki Y, Kikumori K, Murayama E. A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled 14-Week Study of Mirogabalin in Chinese Patients with Diabetic Peripheral Neuropathic Pain. Pain Ther. 2024 Aug;13(4):937-952. doi: 10.1007/s40122-024-00617-2. Epub 2024 Jun 19. PMID 38896199